CLINICAL TRIAL: NCT05468489
Title: A Randomized, Open-label Study of Serplulimab Plus Chemotherapy (Carboplatin-Etoposide) in Comparison With Atezolizumab Plus Chemotherapy in Previously Untreated US Patients With Extensive Stage Small Cell Lung Cancer (ES-SCLC) (ASTRIDE)
Brief Title: To Evaluate Efficacy and Safety of Serplulimab + Chemotherapy (Carboplatin- Etoposide) in US Patients With ES-SCLC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASTRIDE (HLX10-005-SCLC301-E)
Record Dates: First submitted 2022-07-11; First posted 2022-07-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: Extensive Stage Small Cell Lung Cancer; Anti-PD-1 Monoclonal Antibody
MeSH Terms: interventions — Drug Therapy; EC regimen; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Serplulimab + chemotherapy (Experimental): Serplulimab + chemotherapy (carboplatin-etoposide)
  Interventions: Drug: Serplulimab + chemotherapy (carboplatin-etoposide)
- Atezolizumab + chemotherapy (Active Comparator): Atezolizumab + chemotherapy (carboplatin-etoposide)
  Interventions: Drug: Atezolizumab + chemotherapy (carboplatin-etoposide)

INTERVENTIONS:
Drug: Serplulimab + chemotherapy (carboplatin-etoposide) — Drug: Serplulimab is an innovative monoclonal antibody targeting PD-1，developed by Shanghai Henlius Biotech, Inc.
  Drug: carboplatin and etoposide chemotherapeutics
  Arms: Serplulimab + chemotherapy
Drug: Atezolizumab + chemotherapy (carboplatin-etoposide) — Drug: Atezolizumab is a monoclonal antibody targeting PD-L1，developed by Roche Pharma AG.
  Drug: carboplatin and etoposide chemotherapeutics
  Arms: Atezolizumab + chemotherapy

SUMMARY:
This is a randomized, open-label study of Serplulimab plus chemotherapy (Carboplatin-Etoposide) in comparison with Atezolizumab plus chemotherapy in previously untreated US patients with ES-SCLC.

Subjects in this study will be randomized to arm A or B at 1:1 ratio as follows:

* Arm A (Serplulimab): Serplulimab + chemotherapy (carboplatin-etoposide)
* Arm B (control): Atezolizumab + chemotherapy (carboplatin-etoposide)

ELIGIBILITY:
Inclusion Criteria:

Voluntary participation in clinical studies.

Male or female aged ≥ 18 years at the time of signing the ICF.

Histologically or cytologically diagnosed with ES-SCLC (according to the Veterans Administration Lung Study Group staging system).

No prior systemic therapy for ES-SCLC.

At least one measurable lesion as assessed according to RECIST 1.1 within 4 weeks prior to randomization.

Major organs are functioning well.

Every effort should be made to provide tumor tissues for the determination of PD-L1 expression.

An ECOG PS score of 0 or 1.

An expected survival ≥ 12 weeks.

Subjects with prior denosumab use that can and agree to switch to bisphosphonate therapy for bone metastases starting prior to randomization and throughout treatment.

Participant must keep contraception.

Exclusion Criteria:

Histologically or cytologically confirmed mixed SCLC.

Known history of severe allergy to any monoclonal antibody.

Known hypersensitivity to carboplatin or etoposide.

Patients with myocardial infarction within half a year before the first dose of the study drug, poorly controlled arrhythmia.

Pregnant or breastfeeding females.

Patients with a known history of psychotropic drug abuse or drug addiction.

Patients who have other factors that could lead to the early termination of this study based on the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | A period from randomization through death regardless of causality (approximately up to 24 months).
  Overall assessment

SECONDARY OUTCOMES:
ORR | approximately up to 14 months
  Objective response rate
PFS | approximately up to 24 months
  Progression-free survival
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | approximately up to 24 months
  Adverse events are described and graded using the grading categories defined in CTCAE, Version 5.0
Maximum Plasma Concentration (Cmax) | approximately up to 24 months
  The maximum concentration (Cmax) of Serplulimab will be measured
Minimum Plasma Concentration (Cmin) | approximately up to 24 months
  The minimum concentration (Cmin) of Serplulimab will be measured
Average Plasma Concentration (Cavg) | approximately up to 24 months
  The average Plasma Concentration (Cavg) of Serplulimab will be measured

CONTACTS AND LOCATIONS:
Locations (67):
- United States (67):
  - Alabama Oncology, Birmingham, Alabama
  - City of Hope - Phoenix, Goodyear, Arizona
  - Arizona Clinical Research Center (ACRC), Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Compassionate Care Research Group, Fountain Valley, California
  - Providence Medical Foundation, Fullerton, California
  - Los Angeles Cancer Network, Glendale, California
  - OPN - Oncology Physician Network, Los Alamitos, California
  - Kaiser Permanente Research (Southern California), Los Angeles, California
  - UC Davis, Sacramento, California
  - UCHealth Memorial Hospital North, Colorado Springs, Colorado
  - Banner MD Anderson Cancer Center (BMDACC), Greeley, Colorado
  - MD Anderson- North Colorado Medical Center, Greeley, Colorado
  - Advanced Cancer Treatment Centers, Brooksville, Florida
  - Cancer Specialists North Florida, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Affiliates- (Ocala Oncology - Main), Ocala, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - BRCR Global, Plantation, Florida
  - Napa Research, Pompano Beach, Florida
  - Advanced Research, Tamarac, Florida
  - City of Hope- Chicago, Chicago, Illinois
  - Cancer Center of Decatur, Decatur, Illinois
  - Accellacare of Duly, Tinley Park, Illinois
  - Northwest Cancer Centers, Dyer, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Pikeville Hospital, Pikeville, Kentucky
  - CHRISTUS St. Frances Cabrini Cancer Center, Alexandria, Louisiana
  - Pontchartrain Cancer Center, Hammond, Louisiana
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Health Partners Cancer Center at Regions Hospital, Saint Paul, Minnesota
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - North Mississippi Medical Center Hematology and Oncology Clinic, Tupelo, Mississippi
  - MidAmerica Division Inc., c/o Research Medical Center, Kansas City, Missouri
  - Lake Regional, Osage Beach, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Health, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Regional Cancer Care Associates LLC RCCA, Freehold, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Elmhurst (BRANY site), Elmhurst, New York
  - Northwell Health, Lake Success, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Great Lakes Cancer Care (Kaleida Health), Williamsville, New York
  - Summa Health, Akron, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Cancer Center, Canton, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Tricounty Hematology and Oncology Associates, Massillon, Ohio
  - CharterCARE (Roger Williams), Providence, Rhode Island
  - Monument Health, Rapid City, South Dakota
  - CHRISTUS Institute for Innovation & Advanced Clinical Care, Corpus Christi, Texas
  - DHR Research, Edinburg, Texas
  - Millennium Research and Clinical Development, Houston, Texas
  - Lumi Research, Kingwood, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - The University of Texas Health Science Center at Tyler/HOPE Cancer Center, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - American Oncology Network Vista Oncology Division, Olympia, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - West Virginia University Cancer Institute, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Froedtert Hospital- Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No